CLINICAL TRIAL: NCT06600581
Title: Randomized Adaptive Study for Safety and Efficacy of Pluripotent Cell Secretome on Muscle Performance in Seniors With Sarcopenic Obesity
Brief Title: Safety and Efficacy of IMM01-STEM Against Placebo on Muscle Performance in Seniors With Obesity and Muscle Weakness
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STEM-META
Record Dates: First submitted 2024-08-02; First posted 2024-09-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Muscle Performance; Sarcopenic Obesity
Keywords: Muscle Performance; Sarcopenic Obesity
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: STEM-META is a placebo-controlled, randomized, dose expansion study that begins with 4 parallel dosing groups and one placebo control group (phase IIa). The treatment period and follow up will last 16 weeks, then an interim adaptation will initiate the second phase of the study (IIb).
  Treatment Groups
  Group 1 - Placebo - 2 mL USP injectable saline, twice a week Group 2 - 0.5 mg total protein in 2 mL final volume, twice a week Group 3 - 1 mg total protein in 2 mL final volume, once a week, alternating with saline Group 4 - 1 mg total protein in 2 mL final volume twice a week Group 5 - 2 mg total protein in 2 mL final volume, once a week, alternating with saline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The following roles indicated below will not be made aware of the treatment group assignment during the trial:
  Participants Investigators Outcomes assessor
  The person responsible for drug dispensing (pharmacist) will be unblinded
  Sponsor staff or designees may be unblinded to complete ongoing safety oversight and surveillance reporting.
  A planned unblinding will take place at the interim analysis for dose selection in the next phase and futility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (Placebo Comparator): Placebo - 2 mL USP injectable saline, twice a week
  Interventions: Other: Placebo
- Group 2 (Experimental): 0.5 mg total protein in 2 mL final volume, twice a week
  Interventions: Biological: IMM01-STEM
- Group 3 (Experimental): 1 mg total protein in 2 mL final volume, once a week, alternating with placebo (saline)
  Interventions: Biological: IMM01-STEM alternating with placebo (saline)
- Group 4 (Experimental): 1 mg total protein in 2 mL final volume twice a week
  Interventions: Biological: IMM01-STEM
- Group 5 (Experimental): 2 mg total protein in 2 mL final volume, once a week, alternating with placebo (saline)
  Interventions: Biological: IMM01-STEM alternating with placebo (saline)

INTERVENTIONS:
Biological: IMM01-STEM — IMM01-STEM is an allogeneic cell-free secretome product derived from partially differentiated human stem cells derived from a pluripotent embryonic stem cell line that was established from a single donor IVF discarded blastocyst. The cells are cultivated in bioreactors and the product of their secretion is collected, purified and concentrated to a standardized formulation. The secretome contains a mixture of molecules related to immunomodulation, growth, and extracellular matrix remodeling. This intervention is given 2mL twice a week.
  Arms: Group 2; Group 4
Other: Placebo — Saline. This intervention is given 2mL twice a week.
  Other Names: Saline
  Arms: Group 1
Biological: IMM01-STEM alternating with placebo (saline) — This intervention consists of IMM01-STEM given once a week and placebo given one a week. IMM01-STEM is an allogeneic cell-free secretome product derived from partially differentiated human stem cells derived from a pluripotent embryonic stem cell line that was established from a single donor IVF discarded blastocyst. The cells are cultivated in bioreactors and the product of their secretion is collected, purified and concentrated to a standardized formulation. The secretome contains a mixture of molecules related to immunomodulation, growth, and extracellular matrix remodeling.
  Arms: Group 3; Group 5

SUMMARY:
Placebo controlled study for safety and efficacy of IMM01-STEM on muscle performance in seniors with obesity and muscle weakness

DETAILED DESCRIPTION:
This will be a two-phase, placebo-controlled, dose expansion study that begins with 4 parallel dosing groups and one placebo control group (phase IIa). The treatment period and follow up will last 16 weeks, then an interim adaptation will initiate the second phase of the study (IIb). The study will target safety parameters, body composition, and muscle strength and function. Additional metabolic, inflammatory, and muscle-adipose crosstalk markers will be monitored.

During screening, a wearable activity tracker will be assigned to each participant to establish a baseline of daily physical activity.

The treatment will be administered by intramuscular (IM) in a regimen of two injections per week with 2-3 days intervals between injections, for 4 weeks. The dosing groups vary by IMM01-STEM total protein and will be adjusted for identical volumes or equivalent saline volume for placebo. The proposed doses will be 0.5 mg administered twice per week; 1 mg once per week (alternating with a placebo given on the second visit of the week); 1 mg twice per week; and 2 mg once per week (also alternating with placebo).

Each participant will be evaluated at baseline, at the time of treatment administration during the treatment period, then monthly until the end of trial.

Interim analysis with the purpose of design adaptation will be performed after 10 participants from each group have completed treatment. This point will be marked by the date when the final participant to enroll has completed the final treatment on Week 12. This would occur about 16 weeks after the final participant starts treatment.

Statistical analysis will be performed on all recorded outcomes. All participants will continue to be followed-up per protocol for additional 8 weeks.

Post-adaptation, enrollment will be restarted in accordance with the new randomization rules in a 2-arm placebo-controlled study (IIb). The best responding dose will be chosen, or the most convenient treatment (lowest dose, less frequent administration) in the case that all treatment arms responded equally at interim analysis. An amended clinical protocol will be submitted prior initiation of the phase IIb study.

Study participants will sign a written Informed Consent Form (ICF) prior to any study-related procedures. Treatment must begin within 28 days of signing the ICF, during which participant screening and any necessary drug wash-out period must be completed. Screening assessments will be conducted as specified in the Schedule of Activities of the protocol, after which the study participants' eligibility will be determined based on the inclusion and exclusion criteria.

Site staff will administer study medication by IM injection in the gluteal area using a small-gauge needle at all scheduled treatment visits. If gluteal area is not feasible, alternatively i.m. injection can be administered in the quadriceps or deltoid area. After each administration of study medication, participants will be observed for 1 hour to monitor for acute injection-related reactions and other early onset treatment-related AEs.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female
* Age 60 to 80 years of age at the time of signing the informed consent.
* Race/nationality: all races and ethnicities accepted for which there are validated reference values for obesity and sarcopenia diagnostic criteria
* Disease characteristics: To be eligible, the participant must meet at least one criterion for obesity and at least one criterion for sarcopenia, as defined below:

Obesity:

Abdominal obesity defined by a waist circumference ≥ 40 inches (102 cm) for men, ≥ 35 inches (88 cm) for women (American Heart Association) Abdominal obesity as a waist-to-hip ratio of at least 0.90 in men and 0.85 or more for women (World Health Organization)

Sarcopenia:

Grip strength women: < 16 kg, men: < 27 kg in the dominant hand Gait speed < 0.8 m/s (men and women)

Acceptable stages:

STAGE I: No complications attributable to altered body composition and skeletal muscle functional parameters STAGE II: Presence of up to two complications attributable to altered body composition and skeletal muscle functional parameters (e.g. metabolic syndrome components, disabilities resulting from high fat mass and/or low muscle mass, cardiovascular and respiratory disease). Limitations apply (see exclusion criteria).

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the STEM-META clinical protocol
* In order to understand the nature of this study it is expected that most participants will be able to speak, read, and understand English, or Spanish however, additional translations of the informed consent may be made available after study initiation to include additional languages for participants
* Study participant is willing and able to comply with all study requirements, according to the judgment of the Investigator.
* To be eligible for enrollment and for each treatment administration, the vital signs pre-dose, should be in the following ranges. If the vitals are outside of the range, will be reassessed 3 times at 10 minutes resting intervals.

Heart rate >50 and <100 bpm Systolic pressure >100 and <170 mmHg Diastolic pressure >50 and <100 mmHg Blood oxygenation (by pulse-oximetry) >95%

Exclusion Criteria:

* Unmanaged/uncontrolled comorbidities (examples include high blood pressure, hyperglycemia, unstable angina, deep vein thrombosis, hepatic cirrhosis, peptic ulcers, complicated GERD, COPD, asthma etc.) as judged by the investigator.
* Type 1 Diabetes Mellitus, insulin-dependent Type 2 Diabetes mellitus, or hemoglobin A1C level >7.0%
* Severe obesity, or class III obesity (CDC criteria, BMI >40)
* Current diagnosis of major psychiatric disorders that may impact participation, as judged by the investigator.
* Conditions that interfere with gait balance or mobility, such as severe arthritis of lumbo-sacral area, hip or lower extremities if gait speed is used for inclusion criteria
* Conditions that interfere with ability to measure grip strength including hand arthritis, carpal tunnel syndrome and elbow tendinitis if hand grip criteria is used for inclusion
* Study participant has current or past history of invasive malignancy (5 years) excluding non-melanoma skin cancer.
* Inflammatory conditions requiring regular use of oral or parenteral corticosteroids (Raynaud phenomenon, scleroderma, rheumatoid arthritis, LED etc.).
* Cushing's syndrome, Graves disease (hyperthyroidism), or other condition of hormone imbalance caused by genetic or auto-immune disorder. Exceptions include controlled hypothyroidism and polycystic ovarian syndrome.
* Severe cardiovascular disease (including New York Heart Association [NYHA] class III or IV congestive heart failure, clinically significant valvular disease, history of cardiac arrest, presence of an implantable defibrillator)
* Parkinson's disease, multiple sclerosis or other progressive neurological disorders
* Renal disease requiring dialysis, or known renal insufficiency (moderate or severe reduction in GFR≤30 ml/min/1.73 m2)
* Chest pain, severe shortness of breath, or occurrence of other safety concerns during the baseline functional tests
* Study participant is taking or has taken a prohibited medication as defined in Section 6.8.2 of the clinical protocol.
* Participant has had a change in medication to manage comorbid condition(s) (including diabetes, hypertension, asthma, and cardiovascular disease) within 1 month of the Screening visit.
* Weight loss (bariatric) surgery of any type including biliopancreatic diversion with duodenal switch, gastric bypass, sleeve gastrectomy, adjustable gastric banding, 1 year prior enrollment.
* Study participant has previously participated in this study or participant has previously been assigned to treatment in a study of the medication under investigation in this study.
* Study participant has been exposed to an investigational drug or device within 1 year, prior to the first dose of IMP, or is currently participating or planning to participate in another study of an investigational drug.
* Woman of Childbearing Potential (WOCBP) (defined as women with less than 12 months of amenorrhea).
* Unable to understand and/or perform the functional tests, as judged by the Investigator.
* Current physical/rehabilitation therapy (except for passive physical therapy)
* Substance abuse (including but not limited to alcohol, cannabis, narcotics, pain medication) as judged by the investigator.
* Smoking or vaping of products containing nicotine, tobacco or any other products, currently and in the past 1 year.
* Study participant is known positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb) or human immunodeficiency virus-1/2 antibody (human immunovirus 1/2Ab)
* All participants will be encouraged to follow a healthy diet. Caloric restriction will not be pursued.
* Smoking of tobacco, marijuana or any other inhaled products (vaping) are prohibited during treatment and during the follow-up period
* There is no restriction on caffeine consumption
* Occasional alcohol consumption is acceptable, however the participants will be prohibited to consume alcohol 72 hours (3 days) prior medical and laboratory visits
* All participants in the trial (including placebo group) will be encouraged to increase daily physical activities. The participants can follow any preferred physical activity (walking, running, swimming, bicycle, treadmill, etc.), it can be evaluated by summed duration of a variety of activities, such as household work. The activity is measured by the sensors of the wearable activity tracker; thus, the nature of the activity is not critical.
* Activities that are conductive to falls and accidents are discouraged. Examples include horse riding, skiing, skydiving, scuba diving, mountain biking, bungee jumping, etc.
* Participant must be able to wear an activity tracker device daily, optional during sleep, and must be aware of the requirements to charge the tracker or transfer the data.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Time Frame: Day 0 to Day 28
  Safety and tolerability of the IP will be measured by regular monitoring of study subjects' vital signs, blood and urine testing, symptom assessments, physical examinations and physical function testing to identify changes that may be related to the IP. Monitoring begins before treatment and continues for three months following the completion of treatment.
Change over time in gait speed | Time Frame: Day 0 to Day 171
  Muscle strength and function efficacy information from this measure will be used to determine a dosing regimen for a confirmatory expanded study. This will be done using the The European Working Group on Sarcopenia in Older People (EWGSOP2) diagnostic criteria of sarcopenia gait speed.

SECONDARY OUTCOMES:
Change over time in grip strength | Time Frame: Day 0 to Day 171
  Muscle strength and function efficacy information from this measure will be considered for alternative efficacy outcome post interim adaptation. This will be done using the The European Working Group on Sarcopenia in Older People (EWGSOP2) diagnostic criteria of sarcopenia hand grip strength.
Change over time in body composition using DXA | Time Frame: Day 0 to Day 171
  This outcome may be considered for alternative efficacy outcome post interim adaptation.
Change over time in actigraphy parameters as reported by a wearable activity tracker | Time Frame: Day 0 to Day 171
  This purpose of this measurement is to evaluate additional outcomes that may be considered for alternative efficacy outcome post interim adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lane, PhD, Study Director — Chief Science Officer at Immunis, Inc.
Locations (4):
- United States (4):
  - National Institute of Clinical Research (NICR), Garden Grove, California
  - National Institute of Clinical Research (NICR), Pomona, California
  - Johnson Country Clinical Trials (JCCT), Lenexa, Kansas
  - Tekton Research, Wichita, Kansas

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data (IPD) available to other researchers.